CLINICAL TRIAL: NCT05876130
Title: Postoperative Hypofractionated Intensity-modulated Radiotherapy Endometrial Cancer: A Prospective Phase II Trial (POHIM_EM Trial)
Brief Title: Postoperative Hypofractionated Intensity-modulated Radiotherapy Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Park, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-09-123
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Endometrial Cancer
Keywords: radiation therapy; hypofractionation
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: hypofractionated IMRT (2.5 Gy x 16 fractions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- POHIM_EM (Experimental): adjuvant hypofractionated IMRT for endometrial cancer
  Interventions: Radiation: POHIM_EM

INTERVENTIONS:
Radiation: POHIM_EM — hypofractionated intensity-modulated radiation therapy (2.5 Gy/fraction, 16 fractions)

SUMMARY:
To investigate the non-inferiority of disease-free survival in women who received hypofractionated intensity-modulated whole pelvic radiation therapy (2.5 Gy x 16 fractions) after curative surgery for stage III endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed endometrioid type endometrial cancer
* completion of hysterectomy and surgical staging
* pathologically confirmed FIGO stage III
* ECOG performance status 0 or 1
* adjuvant chemotherapy was done or planned

Exclusion Criteria:

* presence of distant metastasis
* previous history of pelvic radiotherapy
* severe and unstable medical condition
* previous history of other carcinoma except for thyroid cancer, skin cancer, and endometrial cancer

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival rate | 5 years
  disease-free survival rate after the time of surgery

SECONDARY OUTCOMES:
acute toxicities | 3 months
  acute toxicities within 3 months according to CTCAE v5.0
late toxicities | 5 years
  late toxicities according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No